CLINICAL TRIAL: NCT00002216
Title: A Comparison of a Four-Drug Regimen Comprised of 141W94, 1592U89, and Combivir With a Three-Drug Regimen Comprised of Nelfinavir and Combivir in Antiretroviral-Naive HIV-Infected Patients.
Brief Title: A Comparison of Two Multi-Drug Therapies in HIV-Infected Patients Who Have Never Received Anti-HIV Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 280C; UNAP 11; NZTA 4002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; abacavir; amprenavir; Nelfinavir

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to compare 2 combination drug therapies in HIV-infected patients who have never received anti-HIV treatment.

DETAILED DESCRIPTION:
In this open-label study antiretroviral-naive patients are randomized to one of two drug regimens:

Arm I: 141W94 (amprenavir), 1592U89 (abacavir), and Combivir (3TC/AZT tablet). Arm II: Nelfinavir and Combivir.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* CD4 count > 50.
* HIV RNA > 5,000.
* No active AIDS (excluding CD4 count < 200).
* Ability to comply with dosing schedule and protocol evaluations.

Prior Medication:

Allowed:

* 3TC or any protease inhibitor, if < 1 week of therapy.
* Other nucleoside analogs, if < 4 weeks of therapy.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active AIDS (not including CD4 count < 200).
* Malabsorption syndrome affecting drug absorption.

Concurrent Medication:

Excluded:

Enrollment in any other investigational drug protocol.

Prior Medication:

Excluded:

Non-nucleoside reverse transcriptase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anderson Clinical Research, Pittsburgh, Pennsylvania, United States